CLINICAL TRIAL: NCT01445821
Title: Randomized Study of Different Non-myeloablative Conditioning Regimens With Hematopoietic Stem Cell Support in Patients With Scleroderma (Autologous Systemic Sclerosis Immune Suppression Trial - II ASSIST-IIb)
Brief Title: Autologous Stem Cell Systemic Sclerosis Immune Suppression Trial
Acronym: DIScl2011
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Developed a better regimen: DIAD. Cast. 2018 NCT03593902
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, Chief, Division of Medicine-Immunotherapy and Autoimmune Diseases; Professor in Medicine-Immunotherapy and Autoimmune Diseases, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASSIST IIb
Record Dates: First submitted 2011-09-29; First posted 2011-10-04 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-06

CONDITIONS: Scleroderma, Systemic
Keywords: Autologous Stem Cell Transplantation
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Cyclophosphamide; Mesna; thymoglobulin; Methylprednisolone; Methylprednisolone Hemisuccinate; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclophosphamide rATG/HSCT (Active Comparator): The control arm will have the same conditioning regimen used in ASSIST study. The conditioning regimen will be 200 mg/kg of intravenous cyclophosphamide given in 4 equal fractions on days -5 through -2 with intravenous mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 and then 1.5 mg/kg from day-4 thru day -1. Methylprednisolone 1000 mg will be used infused intravenously before each dose of rATG. Peripheral blood stem cells (PBSC) will be infused intravenously on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment.
  Interventions: Biological: Peripheral Blood Stem Cells; Drug: Cyclophosphamide; Drug: Mesna; Drug: rATG; Drug: Methylprednisolone; Drug: Filgrastim
- Cyclophosphamide rATG/Fludarabine/HSCT (Experimental): The conditioning regimen will be 120 mg/kg of intravenous cyclophosphamide given in 2 equal fractions on days -3 and -2 with intravenous mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 and then 1.5 mg/kg from day-4 thru day -1. Fludarabine 30 mg/m2 will be given IV on days -5, -4, and -3. Methylprednisolone 1000 mg will be used infused intravenously before each dose of rATG. PBSC will be infused intravenously on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment.
  Interventions: Biological: Peripheral Blood Stem Cells; Drug: Cyclophosphamide; Drug: Mesna; Drug: rATG; Drug: Methylprednisolone; Drug: Filgrastim; Drug: Fludarabine

INTERVENTIONS:
Biological: Peripheral Blood Stem Cells — Mobilized leukapheresis product
Drug: Cyclophosphamide — An alkylating agent which causes prevention of cell division by forming adducts with DNA
  Other Names: Cytoxan; Neosar; Endoxan
Drug: Mesna — Medication used to decrease the risk of hemorrhagic cystitis prophylaxis
  Other Names: Mesnex
Drug: rATG — A predominantly lymphocyte-specific immunosuppressive agent which contains antibodies specific to the antigens commonly found on the surface of T cells
  Other Names: Thymoglobulin
Drug: Methylprednisolone — Steroid
  Other Names: Solu-Medrol
Drug: Filgrastim — Granulocyte-colony stimulating factor (G-CSF); a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  Other Names: Neupogen; G-CSF; Granix; Zarxio
Drug: Fludarabine — Purine analog which inhibits DNA synthesis or repair
  Other Names: Fludara
  Arms: Cyclophosphamide rATG/Fludarabine/HSCT

SUMMARY:
ASSIST I was the first randomized trial in patients with scleroderma to not just slow disease progression but rather actually reverse it. It is the first treatment to have ever demonstrated reversal of lung disease in scleroderma with improvement in FVC, total lung capacity (TLC), high-resolution computed tomography (HRCT), and QOL. We now, therefore, purpose to compare the ASSIST I conditioning regimen of cyclophosphamide and rATG to a less intense regimen of rATG/cyclophosphamide/Fludarabine. In the new regimen the cyclophosphamide dose is decreased to 120mg/kg (60mg/kg/day x 2) compared to 200mg/kg (50mg/kg/day) in the standard regimen. The lower dose of cyclophosphamide will be less cardiotoxic. This study will determine if the less cardiotoxic regimen will be safer than the standard regimen and as effective as the standard regimen.

DETAILED DESCRIPTION:
Mobilization. For patients in both arms undergoing hematopoietic stem cell transplantation (HSCT), peripheral blood stem cells (PBSC) will be mobilized with cyclophosphamide (2 g/m2) followed by 5-10 mcg/kg subcutaneous filgrastrim daily from day 5 until completion of apheresis. Mobilized hematopoietic stem cells (HSC) will be collected by apheresis on day 10 and cryopreserved without selection or manipulation. There will be an interval of at least 17 days between mobilization of PBSC and start of conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 17- 60 years old at the time of pretransplant evaluation
2. An established diagnosis of scleroderma
3. Diffuse cutaneous scleroderma with involvement proximal to the elbow or knee and a Rodnan score (see Appendix V) of > 14 AND

   Scleroderma with any one of the following:
   1. DLCO < 80% of predicted or decrease in lung function (DLCO, DLCO/VA or FVC) of 10% or more over 12 months.
   2. Pulmonary fibrosis or alveolitis on CT scan or chest X-ray (CXR) (ground glass appearance of alveolitis).
   3. Abnormal EKG [non-specific ST-segment and T-wave (ST-T) (pattern in electrocardiogram) wave abnormalities, low QRS (a pattern seen in an electrocardiogram that indicates the pulses in a heart beat and their duration) voltage, or ventricular hypertrophy], or pericardial effusion or pericardial enhancement on MRI
   4. Gastrointestinal tract involvement confirmed on radiological study. Radiologic findings of scleroderma are small bowel radiographs showing thickened folds with dilated loops, segmentation, and flocculation +/- diverticula, or pseudodiverticula. A hide-bound appearance due to valvulae packing i.e. dilated and crowded circular folds may be present. GI involvement may also be confirmed by D-xylose malabsorption, patulous esophagus on HRCT, or esophageal manometry.

   OR
4. As published in New England Journal of Medicine (NEJM), 2006, 345:25 2655-2709. Limited or diffuse Systemic Sclerosis with (SSCL) with lung involvement defined as active alveolitis on Bronchoalveolar Lavage (BAL) or ground-glass opacity on CT, a DLCO < 80% predicted or decrease in lung function (DLCO/VA, DLCO, FVC) of 10% or more in last 12 months.

Exclusion Criteria:

1. Significant end organ damage such as:

   1. Left Ventricular Function (LVEF) < 40% on echocardiogram.
   2. Untreated life-threatening arrhythmia.
   3. Active ischemic heart disease or heart failure.
   4. End-stage lung disease characterized by TLC<45% of predicted value, or DLCO hemoglobin corrected < 30% predicted .
   5. Pulmonary arterial hypertension defined on right heart catheterization as:

      1. a resting Mean Pulmonary Artery Pressure (mPAP) > 25 mmHg;
      2. a mPAP > 30 mmHg following a 500-1000 ml normal saline bolus;
      3. pulmonary vascular resistance (PVR) > 240 dynes*s/cm5 (> 3 Wood units) ; or
      4. a decrease in cardiac output with fluid challenge (500 - 1000 cc Normal Saline (NS) in 10 minutes) If fluid challenge cannot be done because right atrial (RA) pressure > 12mm Hg or pulmonary capillary wedge pressure (PCWP) > 15 m Hg at rest or must be stopped due to safety concerns, patient is excluded as candidate.
   6. Serum creatinine > 1.4 mg/dl.
   7. Liver cirrhosis, transaminases > 3x of normal limits or bilirubin > 2.0 unless due to Gilbert's disease.
   8. Pericardial effusion > 1 cm on cardiac MRI unless successful pericardiocentesis has been performed
   9. Occult or clinical constrictive pericarditis
   10. On echocardiogram tricuspid annular peak systolic excursion (TAPSE) ≤ 1.8 cm or, grade II or worse Right Ventricular (RV) or Left Ventricular (LV) diastolic dysfunction
   11. On cardiac MRI, a diastolic septal bounce or diastolic septal flattering (D-sign), or diffuse myocardial gadolinium enhancement, or diffuse hypokinesis (patchy late gadolinium myocardial enhancement are not exclusion criteria)
   12. Ventricular tachycardia (sustained or non-sustained, multifocal or unifocal) on EKG or 24 hour Holter
2. HIV positive.
3. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.
4. Prior history of malignancy
5. Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
6. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
7. Inability to give informed consent.
8. Major hematological abnormalities such as platelet count < 100,000/ul or absolute neutrophil count (ANC) < 1000/ul.
9. Hepatitis B or C positive

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide rATG/HSCT: Conditioning regimen will be 200 mg/kg of intravenous cyclophosphamide given in 4 equal fractions on days -5 through -2 with IV mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 and then 1.5 mg/kg from day-4 thru day -1. Methylprednisolone 1000 mg will be used infused intravenously before each dose of rATG. Peripheral blood stem cells (PBSC) will be infused intravenously on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment.
  Peripheral Blood Stem Cells: Mobilized leukapheresis product
  Cyclophosphamide: Alkylating agent
  Mesna: Used to decrease the risk of hemorrhagic cystitis
  rATG: Immunosuppressive agent which contains antibodies specific to the antigens
  Methylprednisolone: Steroid
  Filgrastim: Granulocyte-colony stimulating factor (G-CSF); a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells
- Cyclophosphamide rATG/Fludarabine/HSCT: Conditioning regimen will be 120 mg/kg of IV cyclophosphamide given in 2 equal fractions on days -3 and -2 with IV mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 then 1.5 mg/kg from day-4 thru day -1. Fludarabine 30 mg/m2 will be given IV on days -5, -4, and -3. Methylprednisolone 1000 mg will be used infused IV before each dose of rATG. PBSC will be infused IV on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and cont. until neutrophil engraftment.
  Peripheral Blood Stem Cells: Mobilized leukapheresis product
  Cyclophosphamide: Alkylating agent
  Mesna: Used to decrease the risk of hemorrhagic cystitis
  rATG: Immunosuppressive agent which contains antibodies specific to the antigens
  Methylprednisolone: Steroid
  Filgrastim: Granulocyte-colony stimulating factor (G-CSF);glycoprotein that stimulates the bone marrow to produce granulocytes/stem cells
  Fludarabine: Purine analog which inhibits DNA synthesis/repair
Period: Overall Study
Arm/Group | Cyclophosphamide rATG/HSCT | Cyclophosphamide rATG/Fludarabine/HSCT
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cyclophosphamide rATG/HSCT: Conditioning regimen: 200 mg/kg of intravenous cyclophosphamide given in 4 equal fractions on days -5 through -2 with intravenous mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 and then 1.5 mg/kg from day-4 thru day -1. Methylprednisolone 1000 mg will be used infused intravenously before each dose of rATG. Peripheral blood stem cells (PBSC) will be infused intravenously on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment.
  Peripheral Blood Stem Cells: Mobilized leukapheresis product
  Cyclophosphamide: An alkylating agent
  Mesna: Used to decrease the risk of hemorrhagic cystitis
  rATG: Immunosuppressive agent which contains antibodies specific to the antigens
  Methylprednisolone: Steroid
  Filgrastim: Granulocyte-colony stimulating factor (G-CSF); a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells
- Cyclophosphamide rATG/Fludarabine/HSCT: Conditioning regimen: 120 mg/kg of IV cyclophosphamide given in 2 equal fractions on days -3 and -2 with IV mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 and then 1.5 mg/kg from day-4 thru day -1. Fludarabine 30 mg/m2 will be given IV on days -5, -4, and -3. Methylprednisolone 1000 mg will be used infused IV before each dose of rATG. PBSC will be infused IV on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and cont. until neutrophil engraftment.
  Peripheral Blood Stem Cells: Mobilized leukapheresis product
  Cyclophosphamide: Alkylating agent
  Mesna: Used to decrease the risk of hemorrhagic cystitis
  rATG: Immunosuppressive agent which contains antibodies specific to the antigens
  Methylprednisolone: Steroid
  Filgrastim: Granulocyte-colony stimulating factor (G-CSF);glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells
  Fludarabine: Purine analog which inhibits DNA synthesis/repair
- Total: Total of all reporting groups
Arm/Group | Cyclophosphamide rATG/HSCT | Cyclophosphamide rATG/Fludarabine/HSCT | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.8 [23 to 59] | 45.6 [19 to 60] | 44.2 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 17 | 37
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Skin Score Prior to Treatment [Mean (Full Range); unit: units on a scale] — Modified Rodnan Skin Score range from 0 (normal thickness of skin) to 51 (severe thickness of skin)
  units on a scale | 26.1 [13 to 48] | 22.8 [11 to 40] | 24.14 [11 to 48]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure will not occur until a minimum of 12 months after treatment at which time failure is defined as:
  1. Increase of skin score (if > 14 on enrollment) by > 25% above enrollment value and must be documented on 2 occasions at least 6 months apart
  2. Deterioration in percent predicted FVC by 10% below enrollment level, due to systemic sclerosis, and documented on 2 occasion at least 6 months apart
Time Frame: up to and post 12 months of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Cyclophosphamide rATG/Fludarabine/HSCT: Conditioning regimen will be 120 mg/kg of intravenous cyclophosphamide given in 2 equal fractions on days -3 and -2 with intravenous mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 and then 1.5 mg/kg from day-4 thru day -1. Fludarabine 30 mg/m2 will be given IV on days -5, -4, and -3. Methylprednisolone 1000 mg will be used infused intravenously before each dose of rATG. PBSC will be infused intravenously on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment.
  Peripheral Blood Stem Cells: Mobilized leukapheresis product
  Cyclophosphamide: An alkylating agent which causes prevention of cell division by forming adducts with DNA
  Mesna: Medication used to decrease the risk of hemorrhagic cystitis prophylaxis
  rATG: A predominantly lymphocyte-specific immunosuppressive agent which contains antibodies specific to the antigens commonly found on the surface of T cells
  Methylpredni
Arm/Group | Cyclophosphamide rATG/HSCT | Cyclophosphamide rATG/Fludarabine/HSCT
Number analyzed (Participants) | 17 | 15
Participants | 2 | 2

2. Secondary Outcome: Survival of Treatment
Description: Survival of Hematopoietic Stem Cell Transplant.
Time Frame: up to 12 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide rATG/HSCT | Cyclophosphamide rATG/Fludarabine/HSCT
Number analyzed (Participants) | 22 | 22
Participants | 22 | 21

ADVERSE EVENTS:
Time Frame: during treatment at 6 months then yearly for up to 5 years post transplant
Groups:
- Cyclophosphamide rATG/HSCT: Control arm will have the same conditioning regimen used in ASSIST study. The conditioning regimen will be 200 mg/kg of intravenous cyclophosphamide given in 4 equal fractions on days -5 through -2 with intravenous mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5 and then 1.5 mg/kg from day-4 thru day -1. Methylprednisolone 1000 mg will be used infused intravenously before each dose of rATG. Peripheral blood stem cells (PBSC) will be infused intravenously on day 0. Filgrastim 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment.
  Peripheral Blood Stem Cells: Mobilized leukapheresis product
  Cyclophosphamide: An alkylating agent which causes prevention of cell division by forming adducts with DNA
  Mesna: Medication used to decrease the risk of hemorrhagic cystitis prophylaxis
  rATG: A predominantly lymphocyte-specific immunosuppressive agent which contains antibodies specific to the antigens commonl
Arm/Group | Cyclophosphamide rATG/HSCT | Cyclophosphamide rATG/Fludarabine/HSCT
All-Cause Mortality (participants affected / at risk) | 2/22 | 3/22
Serious Adverse Events (participants affected / at risk) | 2/22 | 3/22
Other Adverse Events (participants affected / at risk) | 3/22 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide rATG/HSCT (N=22) | Cyclophosphamide rATG/Fludarabine/HSCT (N=22)
Scleroderma Disease Related (General disorders) | 2 (2) | 3 (3) — Mortality due to disease progression
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide rATG/HSCT (N=22) | Cyclophosphamide rATG/Fludarabine/HSCT (N=22)
Plueral Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pleural Effusion
Disease Related Pericardial Effusion (Cardiac disorders) | 2 (2) | 2 (2) — Scleroderma related pericardial effusion
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 1 (1) — Cardiac Tamponade Requiring Pericardiocentesis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes